CLINICAL TRIAL: NCT00905385
Title: Phase I/II Single-Site, Randomized and Double-Blinded Trial to Further Characterize the HCD50, HCD90 and Transmissibility of Nontypeable Haemophilus Influenzae in a Human Colonization Model in Healthy Adults
Brief Title: Nontypeable H. Influenzae in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 07-0091; H flu Extension
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2010-07

CONDITIONS: Haemophilus Influenzae (NTHI)
Keywords: nontypeable Haemophilus influenzae, NTHi
MeSH Terms: conditions — Haemophilus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Low Dose: 3,200 CFU (Experimental): 5 subjects inoculated with 3,200 colony forming units (CFU).
  Interventions: Biological: NTHi Strain 2019
- High Dose: 32,000 CFU (Experimental): 5 subjects inoculated with 32,000 colony forming units (CFU).
  Interventions: Biological: NTHi Strain 2019

INTERVENTIONS:
Biological: NTHi Strain 2019 — Nontypeable Haemophilus influenzae (NTHi) strain 2019 StrR Number 1 is an antibiotic susceptible clinical strain that has a point mutation in the rRNA that renders the isolate resistant to streptomycin. This agent will be introduced by nasal droplets.

SUMMARY:
The purpose of this study is to learn more about the safety of Haemophilus (H.) influenzae, its ability to produce adverse reactions and to live in the nose and throat. The nose and throat of healthy adults will be populated with a specific type of H. influenzae Nontypeable Haemophilus influenzae (NTHi) 2019 Streptomycin Resistant (StrR) number 1. Researchers will study whether the germ settles in the nose and throat, whether it causes symptoms after it has been placed in the nose, how long the germs last in the nose and throat, and whether the body tries to produce a permanent defense to the germ. Volunteers will receive a lower dose (3,200 germs) or a higher dose (32,000 germs). Active participation will last about 28 days, including a 3 night hospital stay, additional follow-up visits, followed by a 6 month follow-up phone call. Study procedures will include blood samples, saliva samples, several nose washes and throat swabs.

DETAILED DESCRIPTION:
Haemophilus (H.) influenzae continues to be a major human pathogen causing upper and lower respiratory tract diseases ranging from otitis media and sinusitis to invasive pneumonia. The inoculation by nasal droplets proposed in this trial will introduce the organism into the nasal mucosa, the natural host tissue for H. influenzae colonization. It is hypothesized that this inoculum will elicit the typical nasal colonization seen in healthy individuals. To further develop this colonization model, healthy adults devoid of chronic medical conditions that might predispose the subject to invasive disease, will be enrolled. This study is linked to Division of Microbiology and Infectious Diseases (DMID) protocol 04-022. Final safety and reactogenicity data from DMID 04-022, have been collated. This nasal colonization model evaluated 15 volunteers and determined that the model was safe in these individuals and identified a human colonizing dose (HCD) 50 and HCD 90. However, the confidence intervals for these HCD doses were broad. The goals of this study are to further characterize the safety of this trial and to further refine the HCD 50 and 90 doses. This study is a single-site, randomized and blinded study designed to develop a colonization model for Nontypeable Haemophilus influenzae (NTHi). Ten healthy young adults ages 18-54 will be enrolled and inoculated with either 3,200 colony forming units (CFU) or 32,000 CFU of NTHi strain 2019 Streptomycin Resistant (StrR) number 1 and will be followed with nasal wash and throat swabs to determine whether colonization with NTHi 2019 StrR number 1 develops. Subjects that meet enrollment criteria will be admitted to the inpatient clinical research unit to a private room to stay from day 0 thru the morning of day 3 (visits 2-5) to evaluate for reactogenicity after nasal inoculation. During the hospital stay, subjects will remain in respiratory isolation. On day 0, five volunteers will be inoculated at the lower dose, 3,200 CFU, and five will be inoculated with higher dose, 32,000 CFU. After inoculation, primary volunteers will be followed daily for 6 days (visits 2-8, days 0-6) for clinical assessment and culture. Days 4-6, inoculated volunteers will return on a daily basis for a review of reactogenicity parameters, solicitation of adverse events (AEs), a targeted physical exam and pharyngeal swab and nasal wash specimens will be obtained. On day 6, visit 8, after pharyngeal swab and nasal wash samples have been collected and women of child bearing potential have had a urine pregnancy test performed, inoculated volunteers will receive 3 days of levofloxacin to eradicate any potential colonizing study organisms. Participants will return on days 14 and 28 to assess for any AEs, a targeted physical exam will be performed and pharyngeal swab, nasal wash, blood and saliva will be collected. A telephone visit will be performed 6 months after inoculation. A substudy will be performed to evaluate whether casual contact can serve as a mechanism for transmission of NTHi 2019 StrR number 1 from a colonized individual to a casual contact. Three and up to 10 subjects will be recruited to this substudy. They will spend 3-5 hours per day for 6 days with the subject in nonintimate contact and will be followed with nasal wash and throat swabs to determine whether colonization with NTHi 2019 StrR develops. The primary objective of the study is to evaluate the safety and reactogenicity of NTHi Strain 2019 StrR number 1 administered by nasal drop inoculation. The secondary objectives are to: evaluate the frequency and duration of colonization with NTHi strain 2019 StrR number 1 and to establish a human colonizing dose 5

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Inoculated Volunteers:

* Healthy 18-54 years old (male or female) with no chronic medical conditions with the exception of well-controlled hypertension
* Availability for study visits over the next 1 month
* Normal hemoglobin, white blood cell count, creatinine, alanine aminotransferase (ALT), platelet count
* Signed informed consent form
* In good health as determined by medical history and physical exam on the screening evaluation [including heart rate 55-100 beats per minute (bpm); blood pressure: systolic 90-140 mm Hg and diastolic 50-90 mm Hg]. If the subject is a well trained athlete by the judgment of the Principal Investigator (PI), heart rate of 40-100 bpm is acceptable.
* Negative urine pregnancy test for women of childbearing potential
* If the subject is female and of childbearing potential, she agrees to use acceptable contraception and not become pregnant for the duration of the study. (Acceptable contraception includes abstinence, implants, injectables, combined oral contraceptives, effective intrauterine devices, or a vasectomized partner)
* Negative human immunodeficiency virus (HIV) enzyme linked immunosorbent assay (ELISA) for HIV 1 and 2 or indeterminate Western blot or other assay confirming that the serostatus does not reflect HIV infection, negative hepatitis C and hepatitis B serology or other assay confirming that the serostatus does not reflect active hepatitis C virus (HCV) or hepatitis B virus (HBV) infection
* Negative urine protein and glucose by dipstick
* Subjects must be willing to be housed in the clinical research unit for the first 3 nights of the inoculation period.

Inclusion Criteria for Transmissibility Substudy:

* Healthy 18-54 years old (male or female) with no chronic medical conditions with the exception of well-controlled hypertension
* Normal hemoglobin, white blood cell count, creatinine, ALT, platelet count
* Negative HIV ELISA for HIV 1 and 2 or indeterminate Western blot or other assay confirming that the serostatus does not reflect HIV infection, negative hepatitis C and hepatitis B serology or other assay confirming that the serostatus does not reflect active HCV or HBV infection
* Negative urine protein and glucose by dipstick
* Availability for study visits over the next 1 month
* Signed informed consent form
* In good health as determined by medical history and physical exam on the screening evaluation (including heart rate 55-100 bpm; blood pressure: systolic 90-140 mm Hg and diastolic 50-90 mm Hg). If the subject is a well trained athlete by the judgment of the PI, heart rate of 40-100 bpm is acceptable.
* Negative urine pregnancy test for women of childbearing potential
* If the subject is female and of childbearing potential, she agrees to use acceptable contraception and not become pregnant for the duration of the study. (Acceptable contraception includes abstinence, implants, injectables, combined oral contraceptives, effective intrauterine devices, or a vasectomized partner)
* Subjects must be willing to spend 3-5 hours per day for 6 days in nonintimate contact with their paired inoculated contact.

Exclusion Criteria:

Exclusion Criteria for Inoculated Volunteers:

* Acute illness within the week prior to inoculation
* Acute febrile illness (oral temperature greater than or equal to 100.4 degrees Fahrenheit) on the day of inoculation
* Allergic rhinitis requiring therapy in the past year
* Treatment for sinusitis, otitis, chronic bronchitis, pneumonia, bronchospasm or asthma in the past 5 years
* Abnormal gag reflex
* Active drug or alcohol abuse
* Smoking tobacco within the past year
* Average ingestion of more than one alcoholic beverage per day for women or two alcoholic beverages per day for men
* Splenectomy or disease that results in functional asplenism such as sickle cell diseases
* History of malignancy
* Human immunodeficiency virus (HIV) 1 or 2 infection, autoimmune, immunocompromising diseases, diabetes, or chronic renal, hepatic, pulmonary or cardiovascular diseases
* Uncontrolled depression or depression involving institutionalization, history of schizophrenia or psychosis, history of suicide attempt
* Pregnant or lactating woman
* Use of steroids (systemic, inhaled or intranasal) or other medications that can cause immunosuppression within the past 28 days
* American Indian, Native Alaskan or Native Australian heritage (aboriginal)
* Allergy to penicillin, macrolide, cephalosporin or fluoroquinolone antibiotics
* Use of any antibiotic within the past month
* Close contact (household, work or school contact/sexual contacts with, or frequent and/or prolonged exposure to) with persons less than 5 or greater than 55 years old; chronic smokers, Native Americans or other native populations outlined above, or those having HIV infection, cancer, chronic diseases or other illness causing immunosuppression; or having asthma or chronic lung disease. Specifically, child care and health care workers are excluded
* Use of experimental agents or devices within 30 days prior to study or anticipated use of experimental agents or devices within the 6 months of follow up for this study.
* Receipt of blood products or immunoglobulin in the past 6 months
* Any condition that, in the opinion of the investigator, might interfere with study objectives
* Prior participation in nontypeable Haemophilus influenzae colonization studies

Exclusion Criteria for Transmissibility Substudy:

* Acute illness or fever (oral temperature greater than or equal to 100.4 degrees Fahrenheit) within the week prior to inoculation for their paired inoculated contact
* Allergic rhinitis requiring therapy in the past year
* Treatment for sinusitis, otitis, chronic bronchitis, pneumonia, bronchospasm or asthma in the past 5 years
* Abnormal gag reflex
* Active drug or alcohol abuse
* Smoking tobacco within the past year
* Average ingestion of more than one alcoholic beverage per day for women or two alcoholic beverages per day for men
* Splenectomy or disease that results in functional asplenism such as sickle cell diseases
* History of malignancy
* HIV 1 or 2 infection, autoimmune, immunocompromising diseases, diabetes, or chronic renal, hepatic, pulmonary or cardiovascular diseases
* Uncontrolled depression or depression involving institutionalization, history of schizophrenia or psychosis, history of suicide attempt
* Pregnant or lactating woman
* Use of steroids (systemic, inhaled or intranasal) or other medications that can cause immunosuppression within the past 28 days
* American Indian, Native Alaskan or Native Australian heritage (aboriginal)
* Allergy to penicillin, macrolide, cephalosporin or fluoroquinolone antibiotics
* Use of any antibiotic within the past month
* Close contact (household contact/sexual contact with, or frequent and/or prolonged exposure to) with persons less than 5 or greater than 55 years old; chronic smokers, Native Americans or other native populations outlined above, or those having HIV infection, cancer, chronic diseases or other illness causing immunosuppression; or having asthma or chronic lung disease
* Use of experimental agents or devices within 30 days prior to study or anticipated use of experimental agents or devices within the 6 months of follow up for this study
* Any condition that, in the opinion of the investigator, might interfere with study objectives
* Prior participation in nontypeable Haemophilus influenzae colonization studies

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Subjects evaluated for reactogenicity using a standardized illness assessment form. Information on additional unexpected adverse events, new medications and any non-routine medical visits will be assessed. | From day 0 to 28 and at 6 months.

SECONDARY OUTCOMES:
Frequency and duration of colonization with this bacterium in primary subjects. Nasal wash and pharyngeal swab specimens will be obtained for culture of NTHi 2019 StrR number 1. | Days 0, 3, 4, 5, 6, 14, and 28.
Transmission of NTHi 2019 StrR number 1 to close contacts evaluated. | Days 0, 3, 6, 10, 14, and 28.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa - Infectious Disease Clinic, Iowa City, Iowa, United States